CLINICAL TRIAL: NCT03961477
Title: Effect of Interferential Therapy on Pain, Range of Motion and Quality of Life in Patients With Chronic Non-specific Low Back Pain: A Randomized Controlled Trial
Brief Title: Effect of Interferential l Therapy on Low Back Pain
Acronym: [PTREC]
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ahlia University (Other)
Collaborators: Cairo University (Other)
Responsible Party: Principal Investigator, Dr Sayed Tantawy, Professor, Ahlia University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P.T REC/012/001811
Record Dates: First submitted 2019-05-21; First posted 2019-05-23 (Actual); Last update posted 2019-05-23 (Actual); Status verified 2019-05

CONDITIONS: Low Back Pain
Keywords: Low Back Pain,; Interferential Therapy; Quality of Life
MeSH Terms: conditions — Low Back Pain | interventions — Electric Stimulation Therapy; Exercise Therapy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Each subject in both groups was positioned in prone lying and the area to be treated was exposed. The IF group which included 30 subjects received IF. The IF current was increased gradually according the subject's condition with comfortable tingling sensation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- IF group (Active Comparator): Interferential therpapy
  Interventions: Other: Interferential therapy
- Placebo (No Intervention): No intervention

INTERVENTIONS:
Other: Interferential therapy — Exercise therapy
  Other Names: Exercise therapy
  Arms: IF group

SUMMARY:
Background: Chronic non-specific low back pain is defined as unknown mechanical musculoskeletal pain lasting more than 3 months. Electrotherapy is a non-pharmacologic, non-invasive and simple method back pain treatment that is mainly applied using interferential (IF) therapy. The current study was designed to investigate the effect of IF on pain, range of motion, and quality of life in patients with chronic non-specific low back pain. Materials and methods: 61 patients suffered from chronic non-specific low back pain (CNLBP) were randomly assigned to IF group (n=30) and placebo IF (n=31). The entire patient received suggested exercise 3 times per week for 4 weeks. The outcome measures were visual analogue scale (VAS), lumbar range of motion (ROM) in terms of flexion& extension and the Short Form-36 (SF-36) health questionnaire to evaluate the quality of life (QOL).

DETAILED DESCRIPTION:
Participants The study was conducted in outpatient clinics in Cairo University Hospitals. 60 patients (29 males and 31 females) were invited to participate in the current study. Subjects were included in the study if they had LBP of at least three months duration and aged between 25 and 60 years. Patients with spinal pathology (tumor, nerve root, fracture, and compromise), cardiopulmonary conditions, pregnancy, and received physiotherapy in the last eight weeks or any contraindications to the use of electrotherapy were excluded.

ELIGIBILITY:
Inclusion Criteria:

*Subjects were included in the study if they had LBP of at least three months duration * Age between 25 and 60 years.

Exclusion Criteria:

* Patients with spinal pathology (tumor, nerve root, fracture, and compromise),
* Cardiopulmonary conditions
* Pregnancy,
* Received physiotherapy in the last eight weeks
* Any contraindications to the use of electrotherapy were excluded.

Ages: 25 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 61 (Actual)
Dates: Start 2017-12-05 (Actual); Primary Completion 2018-07-11 (Actual); Study Completion 2018-09-23 (Actual)

PRIMARY OUTCOMES:
Visual Analogue Scale (VAS) | 6 months
  The severity of pain was evaluated using a visual analogue scale (VAS). The participants were requested to put a line on the scale perpendicularly that matched to their pain intensity. VAS scores represent the pain intensity as none, mild, moderate, or severe. The accompanying cutoff was used for the pain scale: 0- 4 , no pain; 5- 44, mild pain; 45- 74, moderate pain; and 75-100, severe pain

CONTACTS AND LOCATIONS:
Overall Officials: Sayed A Tantawy, PhD, Study Director — Cairo University
Locations (2):
- Egypt (2):
  - Dr Dalia Kamel, Giza
  - Dr Sayed Tanatwy, Giza